CLINICAL TRIAL: NCT05746494
Title: The Efficacy of Neural Stimulation in Individuals With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Amy Pinkham, PhD, Principal Investigator, The University of Texas at Dallas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-630
Record Dates: First submitted 2023-02-02; First posted 2023-02-27 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia; Schizo Affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will complete active and sham simulation sessions in a randomized, counterbalanced order about one week apart.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active anodal tDCS first, then Sham tDCS (Experimental): Active anodal tDCS (40 minutes; divided into two 20-minutes sessions) followed by behavioral testing; Washout (about 1 week); sham stimulation (40 minutes; divided into two 20-minutes sessions) followed by behavioral testing.
  Interventions: Device: tDCS
- Sham tDCS first, then Active anodal tDCS (Sham Comparator): Sham tDCS (40 minutes; divided into two 20-minutes sessions) followed by behavioral testing; Washout (about 1 week); Active anodal tDCS (40 minutes; divided into two 20-minutes sessions) followed by behavioral testing Intervention.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — active anodal tDCS and sham tDCS

SUMMARY:
The purpose of this study is to understand the relationship between psychotic symptoms and social functioning in individuals with schizophrenia spectrum disorders. Our goal is to determine whether stimulating the brain using transcranial Direct Current Stimulation (tDCS) can improve symptoms and daily functioning.

DETAILED DESCRIPTION:
Paranoid ideation is a common delusion experienced by individuals with schizophrenia spectrum disorders (SSD) that negatively impacts social interactions and quality of life. Therefore, efforts to reduce paranoid thinking via neuromodulation techniques [e.g., transcranial direct current stimulation (tDCS)] are in development, with amygdala-prefrontal cortex (PFC) circuits targeted as critical components of the neural mechanisms underlying paranoia.

This project aims to alleviate paranoia and improve social functioning in individuals with SSD by implementing tDCS to ventrolateral PFC. A double-blind, within-subjects, crossover design will be used to compare the effects of active vs. sham tDCS. Ecological Momentary Assessments (EMA) will also be utilized to quantify any delayed stimulation effects in daily social interactions.

ELIGIBILITY:
Inclusion Criteria:

* Age = 18-64
* Diagnosed with schizophrenia or schizoaffective disorder
* Having current (in the past week) or recent (in the past month) paranoia

Exclusion Criteria:

* Presence or history of a pervasive developmental disorder or mental retardation as defined by IQ < 70
* Presence or history of neurological or medical disorders that contraindicate neural stimulation (e.g. presence or history of epilepsy, seizures, etc.)
* Demonstrating sensory limitations, including uncorrectable visual or hearing impairments that interfere with assessment
* History of electroconvulsive therapy
* Lack of proficiency in English
* Substance use disorder not in remission in the past 6 months
* Any implanted devices such as pace maker, neurostimulator
* Pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Unversity of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan L, Carrico S, Zhu Y, Ackerman RA, Pinkham AE. Transcranial Direct Current Stimulation Improves Paranoia and Social Functioning in Schizophrenia: A Randomized Clinical Trial. Biol Psychiatry. 2025 Jul 15;98(2):135-143. doi: 10.1016/j.biopsych.2025.01.011. Epub 2025 Jan 22. PMID 39855408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 participants were enrolled and eventually completing the whole procedure.
Period: Overall Study
Arm/Group | Active Anodal tDCS First, Then Sham tDCS | Sham tDCS First, Then Active Anodal tDCS
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Anodal tDCS First, Then Sham tDCS | Sham tDCS First, Then Active Anodal tDCS | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.08 (10.24) | 45.46 (11.30) | 44.74 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 23 | 46
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 13 | 27
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50
Handedness [Number; unit: participants]
  right-handed | 23 | 22 | 45
  left-handed | 3 | 2 | 5
Years of education [Mean (Standard Deviation); unit: years] | 12.42 (2.08) | 13.31 (2.26) | 12.85 (2.20)
The Wide Range Achievement Test-Reading recognition subtest 4 (WRAT-4) [Mean (Standard Deviation); unit: units on a scale] — This scale measures the Intelligence Quotient (IQ). A total final standardized score (adjusted by age) is computed. The range of this total score is from 55 to 145. A higher total score indicates a higher IQ and suggests that the participant is more intelligent.
  units on a scale | 96.11 (9.76) | 94.08 (15.02) | 95.14 (12.47)
Chlorpromazine (CPZ)-equivalent [Mean (Standard Deviation); unit: mg] — This measures the dosage of antipsychotic medications that the participant is taking. A total final score is computed. The range of this total score is from 0 to unlimited. A higher score indicates a higher dosage of antipsychotic medications.
  mg | 468.63 (1150.45) | 396.32 (520.71) | 433.92 (896.59)
Diagnoses [Number; unit: participants] — Two types of diagnoses were included in this study, including schizophrenia (SCZ) and schizoaffective disorder (SCZ-A). Diagnoses were determined via Mini International Neuropsychiatric Interview (MINI) and Structured Clinical Interview for DSM Disorders-Psychosis Module (SCID-P).
  participants
    SCZ | 8 | 13 | 21
    SCZ-A | 18 | 11 | 29
Current/recent paranoia [Number; unit: participants]
  Current | 21 | 17 | 38
  Recent | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: The State Social Paranoia Scale (SSPS)
Description: Paranoid ideation was measured by the State Social Paranoia Scale (SSPS). Participants indicated how much they agree with each of 20 statements (e.g., "Someone was hostile towards me", "Someone was trying to isolate me") using a 5-point Likert scale (1 = do not agree, 5 = totally agree). Scores range from 20-100, and higher scores represent higher state paranoid ideation.
Time Frame: The assessment was completed before the stimulation and 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: The change score of SSPS (pre - post)
Groups:
- Active Visit: Performance at the active visit
- Sham Visit: Performance at the sham visit
Arm/Group | Active Visit | Sham Visit
Number analyzed (Participants) | 50 | 50
The change score of SSPS (pre - post) | 9.72 (14.61) | 3.90 (11.56)
Statistical Analysis 1: Comparison: Active Visit vs Sham Visit; Test type: Other — Omnibus analysis; p = 0.023, ANOVA

2. Primary Outcome: Ecological Momentary Assessment (EMA)-Based Paranoia
Description: Paranoid ideation was measured by Ecological Momentary Assessment (EMA), which involved questions about feelings of paranoia in daily life. The paranoia-related question is as follows: "Since the past alarm, how much have you had thoughts that you really can't trust other people?" The score for this item ranges from 1 to 7, with a higher score indicating a higher level of paranoid thinking.
Time Frame: Change in daily paranoia feelings was assessed from the pre-stimulation EMA period (7 days before the stimulation visit) to the post-stimulation EMA period (7 days after the stimulation visit)
Population: Only 47 (out of 50) participants completed this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EMA-baseline: EMA-baseline
- EMA-active: EMA-active
- EMA-sham: EMA-sham
Arm/Group | EMA-baseline | EMA-active | EMA-sham
Number analyzed (Participants) | 47 | 47 | 47
units on a scale | 3.78 (1.72) | 3.61 (0.91) | 3.96 (1.85)
Statistical Analysis 1: Comparison: EMA-baseline vs EMA-active vs EMA-sham; Test type: Other — Omnibus analysis; p = 0.042, Multilevel Modeling

3. Primary Outcome: Birchwood Social Functioning Scale (SFS)
Description: Social functioning was measured by the Birchwood Social Functioning Scale (SFS). This scale measures social adjustment based on self-reports (4- or 5-point scales), with higher total scores indicating better social functioning (range = 0-223).
Time Frame: The assessment was completed 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Visit | Sham Visit
Number analyzed (Participants) | 50 | 50
units on a scale | 114.21 (22.35) | 114.59 (27.54)
Statistical Analysis 1: Comparison: Active Visit vs Sham Visit; Test type: Other — Omnibus analysis; p = 0.980, t-test, 2 sided

4. Primary Outcome: Ecological Momentary Assessment (EMA)-Based Social Functioning
Description: Social functioning was measured by Ecological Momentary Assessment (EMA) (i.e., questions about daily interactions with others). Two subscores were generated: social interaction frequency (score ranges from 0-5, a higher score indicates more frequent social interactions), social interaction motivation and experience (scores range from 1-7, a higher score indicates higher motivations to interact with others and better experiences during these interactions).
Time Frame: Change in daily interactions was assessed from the pre-stimulation EMA period (7 days before the stimulation visit) to the post-stimulation EMA period (7 days after the stimulation visit)
Population: Only 47 (out of 50) participants completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMA-baseline | EMA-active | EMA-sham
Number analyzed (Participants) | 47 | 47 | 47
score on a scale
  Social interaction frequency | 0.97 (0.76) | 0.91 (0.83) | 0.92 (0.90)
  Social interaction motivation and experience | 3.74 (1.62) | 4.08 (1.68) | 3.71 (1.62)
Statistical Analysis 1: Comparison: EMA-baseline vs EMA-active vs EMA-sham; Test type: Other — Omnibus analysis; p = 0.010, Multilevel Modeling

5. Secondary Outcome: The Trustworthiness Task
Description: Paranoid ideation was measured by the Trustworthiness Task. This task requires participants to indicate how much they trust each of 60 grayscale facial stimuli along a 7-point Likert scale (-3 = very untrustworthy, 3 = very trustworthy). Total scores were calculated by averaging across responses and hence varied from -3 to +3, with higher values indicating a greater tendency to trust others.
Time Frame: The assessment was completed 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Visit | Sham Visit
Number analyzed (Participants) | 50 | 50
score on a scale | 0.07 (1.16) | -0.18 (0.99)
Statistical Analysis 1: Comparison: Active Visit vs Sham Visit; Test type: Other — Omnibus analysis; p = 0.064, t-test, 2 sided

6. Secondary Outcome: The Scrambled-sentences Task (SST)
Description: Paranoid ideation was measured by the Scrambled-sentences task (SST). This task measures the level of paranoia by asking participants to create sentences of either paranoid or nonparanoid meanings, with a greater percentage indicating a higher level of paranoid interpretation bias (range = 0-1).
Time Frame: The assessment was completed 30 minutes after completion of the active/sham stimulation
Population: Only 49 (out of 50) participants completed this task.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Visit | Sham Visit
Number analyzed (Participants) | 49 | 49
score on a scale | 0.46 (0.29) | 0.49 (0.28)
Statistical Analysis 1: Comparison: Active Visit vs Sham Visit; Test type: Other — Omnibus analysis; p = 0.306, t-test, 2 sided

7. Secondary Outcome: The Ambiguous Intentions Hostility Questionnaire (AIHQ)
Description: Paranoid ideation was measured by the Ambiguous Intentions Hostility Questionnaire (AIHQ). Three subscores were generated: AIHQ (blame) (ranging from 3-16, with a higher score indicating a higher level of blaming tendency), AIHQ (hostility) (ranging from 1-5, with a higher score indicating a higher level of hostility), AIHQ (aggression) (ranging from 1-5, with a higher score indicating a higher level of aggression).
Time Frame: The assessment was completed 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Visit | Sham Visit
Number analyzed (Participants) | 50 | 50
score on a scale
  AIHQ (blame) | 8.28 (3.07) | 8.89 (3.22)
  AIHQ (hostility) | 2.09 (0.75) | 2.35 (0.78)
  AIHQ (aggression) | 1.75 (0.40) | 1.78 (0.39)
Statistical Analysis 1: Comparison: Active Visit vs Sham Visit; Test type: Other — Omnibus analysis; p = 0.041, t-test, 2 sided

8. Secondary Outcome: The Hostility Scale of the Personality Inventory for DSM-5 (PID-5-HS)
Description: Paranoid ideation was measured by the Hostility Scale of the Personality Inventory for DSM-5 (PID-5-HS). PID-5-HS contains 10 self-report items assessing pathological hostility. A total score (range from 0-30) was generated to reflect overall hostility level, with higher total scores indicating more hostility.
Time Frame: The assessment was completed 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Visit | Sham Visit
Number analyzed (Participants) | 50 | 50
score on a scale | 9.42 (7.56) | 11.30 (7.57)
Statistical Analysis 1: Comparison: Active Visit vs Sham Visit; Test type: Other — Omnibus analysis; p = 0.019, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Immediately after the stimulation visit, up to 24 hours
Groups:
- Active Visit: Active anodal tDCS (40 minutes; divided into two 20-minutes sessions) followed by behavioral testing
- Sham Visit: Sham tDCS (40 minutes; divided into two 20-minutes sessions) followed by behavioral testing
Arm/Group | Active Visit | Sham Visit
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
The inherent limitations of the assessment tools for measuring social functioning in the lab may have impacted the findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT05746494/Prot_SAP_000.pdf